CLINICAL TRIAL: NCT05837949
Title: Multiple Sclerosis Falls Insight Track: A Personal Health Library to Reduce Falls in Patients With Multiple Sclerosis
Brief Title: Multiple Sclerosis Falls Insight Track
Acronym: MS FIT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Library of Medicine (NLM) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22-36680; 5R01LM013396-02 (NIH)
Record Dates: First submitted 2023-04-17; First posted 2023-05-01 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; Falls; Falling; Closed-loop; Digital health; Falls tracking; Falls prevention; FitBit; Wearables
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: All participants will be given the MS FIT tool intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MS FIT: Falls Insight Track (Experimental): Participants in this arm will receive 12 months use of MS FIT mobile tool intervention
  Interventions: Behavioral: MS FIT: Falls Insight Track

INTERVENTIONS:
Behavioral: MS FIT: Falls Insight Track — Participants will respond to a set of surveys every two weeks to increase communication on falls with their clinician.

SUMMARY:
The purpose of this study is to develop an application: MS Falls Insight Track (MS FIT) which allows patients to log their falls and near falls, view their MS relevant data and responses to the clinic intake survey as well as communicate with their care team about falls and receive educational material on falls prevention.

DETAILED DESCRIPTION:
Falls occur in >50% patients with multiple sclerosis (MS), worsen participation in daily life and increase healthcare costs. To date there are no established, accessible, tools to evaluate and reduce fall risk. MS Falls InsightTrack is a live personal health library that combines a patient's falls-relevant clinical indicators (from the electronic health record, EHR) with patient-generated data (PGD) from commercial wearable tools and patient-reported outcomes (PROs) and community-level data (sociodemographic data from University of California, San Francisco (UCSF) Health Atlas combined with MS-specific resources from the National MS Society). The tool will track falls/near-falls in real- time and report changes in status that require intervention. It will offer customized action prompts to support fall reduction through a behaviorally informed approach. It will be accessed in the clinic and in the patient's home.

Technological features. The tool will be accessible, extensible and scalable. The investigators will use modern technologies and industry standards (e.g back-end: Python, flask framework, PostgreSQL; front-end: HTML, CSS, JavaScript and d3.js). The tool will launch from Epic via SMART on FHIR, and will communicate with patients using MyChart.

Qualifications of team and setting. The UCSF MS Center is a leading clinical research center in the digital space. Our sub-leads are experts in all aspects of the study (digital technology, human-centered design, implementation science, health literacy) with a varied and experienced Stakeholder Advisory Group.

Scientific plan. In Aim 1 (design), the investigators will use a Human-Centered Design approach, engaging 20 patients with MS, clinicians and stakeholders in a series of focus groups, to identify the critical data, devices, visualizations, resources, workflows and accessibility/digital divide considerations for the tool, and the key interventions likely to promote the COM-B model of behavioral change to reduce fall risk.

Our key outcomes will be perceived effectiveness, ease of use and likability. In Aim 2 (evaluate feasibility), investigators will deploy MS Falls Insight Track in 100 diverse adults with MS who are at risk for falls. Participants will wear a Fitbit. The tool will be used by patients in their homes and by clinicians during clinical encounters. The investigators will use an implementation science approach. Our key outcomes will be study retention, tool uptake and sustained use. The investigators will explore impact on fall risk. In Aim 3 (test generalizability) investigators will conduct focus groups with patients with other conditions where falls are common (Orthopedics, Parkinson's Disease, Geriatrics) to understand additional data and design features required to promote generalizability. Our key outcomes will parallel those in Aim 1.

Innovation and Broader Significance. MS Falls Insight Track is a unique, comprehensive, accessible personal health library that can be deployed in larger efficacy trials for falls reduction. Beyond this clinical use case, the closed-loop approach of delivering PGD to the care system and back to the patient, interpreted and actionable, using scalable technology, represents a significant innovation that can sequentially expand the number of wearables, conditions and clinics in which patients and clinical investigators can ask their own questions of PGD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS (relapsing or progressive) by 2017 McDonald Criteria18
* Ages 18 and above
* Any MS therapy, or no treatment
* California resident to enable clinical telemedicine visits if warranted during the study visit
* EDSS 2.0-8.0 (moderate to severe impairment, 7= wheelchair but independent transfers)
* Fall risk, based on MSWS-12 score and previous report of a fall (Hopkins grade ≥1)
* Technological criteria: availability of Wi-Fi in the home or workspace for connectivity.

Exclusion Criteria:

* Cognitive dexterity or visual impairment that, in the opinion of the study neurologist (RB), would put the participant at risk or limit their ability to comply with the study protocol
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients initially use the tool (Adoption) | 6 months
  This will be measured by calculating the percentage of patients who use the tool during the initial month of the study, and by the percentage of patient-clinical dyads who use the tool during the clinical visit
Percentage of patient-clinician encounters initially use the tool (Adoption) | 6 months
  This will be measured by calculating the percentage of patient-clinical dyads who use the tool during the clinical visit.
Percentage of patients who continue to use the tool (Engagement) | 12 months
  This will calculate the percentage of patients who continued to use the patient-facing tool at least quarterly
Percentage of patient-clinician encounters use the tool during the 12-month visit (Engagement) | 12 months
  This will be calculated by the percentage of the clinician-patient dyads in Arm 1 who use the in-visit dashboard at the 12-month clinical visit.
Percentage of patients who respond to fall prompts (Adherence) | 12 months
  Adherence will be measured by the percentage of falls reporting prompts adhered to per participant, as well as percentage of participants adhering to >75% falls prompts

CONTACTS AND LOCATIONS:
Overall Officials: Riley Bove, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The deidentified dataset will be shared with qualified collaborators upon request, provision of CITI and other certifications, and data sharing agreement. We will share the results, once the data are complete and analyzed, with the scientific community and patient/clinician participants through abstracts, presentations and manuscripts.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months post trial
Access Criteria: Qualified collaborators upon request, provision of CITI and other certifications, and data sharing agreement

REFERENCES:
- [Derived] Block VJ, Koshal K, Wijangco J, Miller N, Sara N, Henderson K, Reihm J, Gopal A, Mohan SD, Gelfand JM, Guo CY, Oommen L, Nylander A, Rowson JA, Brown E, Sanders S, Rankin K, Lyles CR, Sim I, Bove R. A Closed-Loop Falls Monitoring and Prevention App for Multiple Sclerosis Clinical Practice: Human-Centered Design of the Multiple Sclerosis Falls InsightTrack. JMIR Hum Factors. 2024 Jan 11;11:e49331. doi: 10.2196/49331. PMID 38206662